CLINICAL TRIAL: NCT05914519
Title: Outcomes and Efficacy of Ejaculatory Preserving Transurethral Resection of Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Sabri Mahmoud, Principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-23-06-02MD
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Ejaculatory Dysfunction; BPH
MeSH Terms: conditions — Ejaculatory Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Procedure: Ejaculatory Preserving Transurethral resection of prostate
- Group 2 (Active Comparator)
  Interventions: Procedure: Standard Transurethral Resection of prostate

INTERVENTIONS:
Procedure: Ejaculatory Preserving Transurethral resection of prostate — Transurethral resection of prostate with preservation of 1cm safety area above verumontanum and without paracollicular digging
  Other Names: EpTURP
  Arms: Group 1
Procedure: Standard Transurethral Resection of prostate — Transurethral resection of prostate including whole adenoma till the capsule.
  Other Names: Standard TURP
  Arms: Group 2

SUMMARY:
The purpose of this study is to assess the outcomes and efficacy of ejaculatory preserving TURP in terms of voiding, erectile function, and ejaculation.

DETAILED DESCRIPTION:
The prostatic gland plays a central role in andrology. It is involved both in fertility and in sexuality with a major role in ejaculation and possibly in orgasm. This could explain the association between the andrological symptoms and prostatic disorders.

The prevalence of Benign Prostatic Hyperplasia (BPH) is approximately 50% for men in their fifties and reaches up to 80% for men over 80 years of age, representing one of the most common diseases affecting males, with potentially significant impact on their quality of life.

It is estimated that around half of men suffering severe or medical treatment unresponsive lower urinary tract symptoms (LUTS) will be offered a surgical procedure to relieve benign prostatic obstruction (BPO).

Despite continuing development of new minimally invasive surgical methods, transurethral resection of the prostate (TURP) still remains the gold standard surgical treatment for LUTS due to BPH.

Although it is benign, this disease has been shown to have a negative impact on the patient's health-related quality of life (HRQL), marked by obstructive and irritative LUTS.

As BPH in most cases is not a life-threatening condition, the main outcomes of its treatment are not only the improvement in LUTS and functional parameters but also quality of life after surgery.

Whilst efficacy of the conventional TURP is proven, a common potentially bothersome side effect, the retrograde ejaculation (RE) which occurs in 65-90% of patients undergoing TURP.

It has been reported that ablative techniques like TURP and recent laser procedures including holmium, thulium and greenlight cause similar rates of ejaculatory dysfunction, occurring in almost three out of four to five men.

For decades, men have been counseled to expect dry orgasm after TURP because of the retrograde flow of semen as a result of bladder neck disruption.

Erectile dysfunction and Ejaculatory dysfunction (EjD) can have a substantial deleterious effect on the Quality of life (QoL) of men who have previously maintained regular sexual activity, inducing significantly increased levels of anxiety and depression.

More recently, a better understanding of ejaculation physiology has enabled the emergence of modified surgical techniques with the aim of preserving antegrade ejaculation.

The key point of standard TURP is resecting the tissues enveloped in the prostatic capsule and the bladder neck, while protecting the urethral tissues below the verumontanum.

The bladder neck plays a significant role in reproduction. For men, bladder neck closure facilitates anterograde ejaculation. It actively contracts the bladder neck during ejaculation through a rich noradrenergic innervation by sympathetic nerves.

Vernet et al. showed that contraction of the bladder neck was not important for anterograde ejaculation. Using endorectal ultrasound videos performed during masturbation in 30 men, it was possible to visualize the bladder neck, the prostate, and the bulbar urethra during ejaculation. They observed that during ejaculation, the verumontanum underwent a slight caudal shift, momentarily making contact with the opposite urethral wall and sperm emitted from the ejaculatory ducts was directed distally by contractions of the external sphincter coordinated with contractions of the bulbar urethra, thus demonstrating the importance of the muscular tissue around the verumontanum and particularly its proximal part. They described this area as a "high-pressure ejaculatory area". The closure of the bladder neck did not seem to play a role in this mechanism. As a result, one can conclude that as long as the tissues around the verumontanum are not injured, ejaculation should still occur even with a well-open bladder neck.

Recently, together with a better understanding of the mechanisms of ejaculation, a greater importance has been given to the impact of dry ejaculation on patients' QoL. A balance between symptomatic improvement in LUTS and preservation of sexual function needs to be addressed for men seeking surgical treatment.

Modifications based on Supramontanal sparing hypothesis have reported favorable outcomes to as high as 92%.

Although preservation of bladder neck structures is often associated with preservation of antegrade ejaculation, the current modern approach is the preservation of the precollicular and para-collicular tissue in the area where the ejaculatory ducts emerge near the verumontanum in the distal apical tissue in laser, aquablation, and bipolar electrosurgical prostatectomy techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 45 years old.
* Drug refractory urinary retention.
* Prostate volume range: 20-60 mL.
* IPSS > 19 after the medical therapy failure.
* Qmax < 10 mL/s.
* PSA < 4 ng/mL.
* Active and healthy sexual life.

Exclusion Criteria:

* History of prostate or urethral surgery.
* Neurogenic bladder.
* UTI.
* Urethral stricture disease.
* prostate cancer.
* Bleeding diathesis.
* Capsular or bladder perforation during surgery.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 103 patients were assessed for eligibility; 8 patients did not meet the criteria and 5 patients refused to participate in the study. The remaining patients were randomly allocated into two equal groups (45 patients in each). All allocated patients were followed-up and analyzed statistically.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 45 | 45
Completed | 43 | 41
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.76 (8.16) | 65.58 (7.98) | 64.17 (8.07)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 45 | 45 | 90
Maximum Flow Rate (Qmax) [Mean (Standard Deviation); unit: ml/sec] — The maximum flow of urine measured by uroflowmetry
  ml/sec | 4.92 (1.73) | 4.5 (1.88) | 4.71 (1.805)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Preservation of Ejaculation
Description: The number of patients who can ejaculate after TURP
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: ejaculatory preserving TURP
- Group 2: classic TURP
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 43 | 41
Participants | 34 | 8

2. Secondary Outcome: Maximum Flow Rate (Qmax)
Description: The maximum flow of urine measured by Uroflowmetry
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 43 | 41
ml/sec | 18.78 (5.16) | 19.71 (6.22)

ADVERSE EVENTS:
Time Frame: 6 months
Description: TURP is an elective surgery that the patient is prepared with full lab and surgical fitness in preoperative assessment furthermore, TURP has a high safety profile that all adverse events rarely lead to mortality
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/45
Other Adverse Events (participants affected / at risk) | 12/45 | 23/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=45) | Group 2 (N=45)
intraperitoneal bladder perforation (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=45) | Group 2 (N=45)
sever irritative LUTS (Renal and urinary disorders) | 4 (9) | 7 (9)
Minor Capsular perforation (Renal and urinary disorders) | 1 | 2
Blood transfusion (Blood and lymphatic system disorders) | 1 | 2
Clot retention (Renal and urinary disorders) | 2 | 4
Stress incontinence (Renal and urinary disorders) | 1 | 2
Bladder neck contracture (Renal and urinary disorders) | 2 | 4
Stricture bulbar urethra (Renal and urinary disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
* Single center study that may result in different findings than elsewhere.
* Small sample size that may produce insignificant results.
* Relatively short period of follow-up.
* We didn't compare Ejaculatory preserving TURP with other established surgical or minimally invasive techniques such as aquablation and Holmium laser enucleation with ejaculatory sparing modifications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT05914519/Prot_SAP_000.pdf